CLINICAL TRIAL: NCT06490432
Title: Pattern of Cardiac Arrhythmia in Patients With Metabolic Dysfunction -Assocatied Steatotic Liver Disease in Sohag University Hospital.
Brief Title: Pattern of Cardiac Arrhythmia in Patients With MASLD
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Rashwan Ahmed, Principal investigator, Sohag University
Other Study IDs: Soh-Med-24-06-04MS
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrhythmia; Metabolic Dysfunction Associated Steatotic Liver Disease
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transient elastography — Device that measures stiffness of liver tissue
  Other Names: Echocardiograpy; ECG

SUMMARY:
Study the relationship between patients with MASLD and cardiac arrhythmia that could be occur in thos patients

DETAILED DESCRIPTION:
Study the cardiac arrhythmia that could be occur in patients suffering form metabolic dysfunction -assocatied steatotic liver disease and risk factors of them

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18years or older Patients with metabolic dysfunction -assocatied steatotic liver disease

Exclusion Criteria:

* RHD Structural heart diseases Liver diseases other than MASLD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study relationship between patients with metabolic dysfunction -assocatied steatotic liver disease and cardiac arrhythmia in those patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Cardiac arrhythmia and MASLD patients | 1 year
  Study metabolic dysfunction -assocatied steatotic liver disease
Cardiac arrhythmia | 1 year
  Study pattern of cardiac arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Mostafa, Lecturer, Study Director — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, So, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee HH, Lee HA, Kim EJ, Kim HY, Kim HC, Ahn SH, Lee H, Kim SU. Metabolic dysfunction-associated steatotic liver disease and risk of cardiovascular disease. Gut. 2024 Feb 23;73(3):533-540. doi: 10.1136/gutjnl-2023-331003. PMID 37907259